# **Informed Consent Form**

**Study Title:** Using the Arts as a Proactive Mental Health Strategy for Generation Z

**Date:** August 31<sup>st</sup>, 2020

#### **FSU CONSENT FORM**

#### Introduction

You are invited to participate in a research study of a technology-based approach for stress- and anxiety-reducing techniques to determine if there is a trained biofeedback response. You were selected as a possible participant because you are a full-time FSU student between the ages of 18 and 24 that is a non-smoker. We ask that you read this form and ask any questions you may have before agreeing to be in the study.

This study is being conducted by Principal Investigators Dr. Theresa van Lith of the Department of Art Education, Dr. Gregg Stanwood of the Department of Biomedical Sciences, and Dr. Scott Pickett of the Department of Behavioral Sciences and Social Medicine. The research coordinator of this study is Andrea Cheshure, MS in Psychology. This study is funded by the National Endowment of the Arts (NEA).

## **Study Purpose**

The purpose of the study is to determine the stress- and anxiety-reducing benefits of a technology-based mental health program for full-time university students over the course of a 5-week period. This will be determined based on the fluctuations in the stress hormone: cortisol. It involves self-care challenges to be completed twice a week that have been developed by a professional art therapist. The study hopes to confirm that there is a biofeedback response to practicing these challenges persistently over the 5 weeks.

#### **Study Procedures**

If you agree to participate in this study, you will be asked to complete two 1-hour meetings on campus, one to be held on the first week of the study and one on the 5<sup>th</sup> week, in addition to participate in self-care challenges twice a week remotely via the Canvas app. These self-care challenges are brief, requiring approximately 15 minutes each and involve practicing techniques for reducing stress and symptoms of anxiety. You would also be committing to providing a total of three passive drool saliva samples (on week 1 and twice on week 5) and completing two self-assessments online. There are two brief self-reporting assessments you will complete through the duration of the study, with each self-care challenge.

# **Risks of Study Participation**

Research studies may involve different kinds and levels of risks or discomforts. These could be physical, emotional, social, economic or legal risks. For this study, the potential risks and discomforts that we know about are described below.

Covid-19. Participants are required to complete two brief in-person sessions with the research coordinator. The research coordinator will be wearing appropriate protective gear and will provide participants with PPE upon entering the building if necessary. Masks will be worn throughout the session, except during the collection of the saliva sample. We have taken the necessary precautions to ensure that risk of exposure is

minimized. If you or anyone you know has been exposed to the virus, or have tested positive in the last 14 days, we ask that you disclose and reschedule your appointment.

Identification through deductive disclosure. That is, there is very unlikely possibility that an individual who is not a part of the research team may accidently gain access to your data (e.g. email address) and be able to identify your responses. However, we have taken several steps in making sure this does not happen including: the use of a person specific code, the data will be kept in a password locked account on Qualtrics.com, and any data that is downloaded by the researchers will be kept on a password protected computer. In the case of presenting data in a professional paper or presentation all data will be presented as aggregate, so no one person will be identifiable.

Please note that Qualtrics has specific privacy policies of its own. If you have concerns, you should consult Qualtrics directly at https://www.qualtrics.com/privacy-statement/.

#### **Benefits**

The potential benefits to study participation are experiencing a decrease in your stress and symptoms of anxiety, as well as learning simple techniques for stress and anxiety reduction that you can use on your own.

#### Cost

There is no cost to you for participating in this study.

#### Compensation

Upon full participation and completion of the study, you will be compensated for your time and inconvenience in the form of a \$10 Amazon gift card. You will also have your name added to a raffle with other study participants for the chance to win one of four \$25 Amazon gift cards.

#### Confidentiality

The records of this study will be kept private and confidential, to the extent allowed by law. In any publications or presentations, we will not include any information that will make it possible to identify you as a subject. Your record for the study may, however, by reviewed by departments at the University with appropriate regulatory oversight. Data collected throughout the study including assessment results, biospecimens, survey responses, and photographs of artwork may be used for scientific and educational purposes. Scientific purposes include storage and maintenance of biospecimens, as well as secondary use of data in future research. Educational purposes include training, supervision, research, and publication. All photographs will be presented in a respectful and professional manner. No information will be recorded in participants' medical record

### **Protected Health Information (PHI):**

Your PHI created or received for the purposes of this study is protected under the federal regulation known as HIPAA. Refer to the HIPAA authorization for details concerning the use of this information.

# **Voluntary Nature of the Study**

Participation in this study is voluntary. Your decision to participate in this study will not affect your current or future relations with the University. If you decide to participate, you are free to withdraw at any time without affecting those relationships.

### **Contacts and Questions**

The researcher facilitating this study is Andrea Cheshure. You may ask any questions you have now, or if you have questions later, you are encouraged to contact her at <a href="mailto:acheshure@fsu.edu">acheshure@fsu.edu</a> or (. You may also contact the Principal Investigators, Dr. Theresa Van Lith at (850) 645-9890, and Dr. Gregg Stanwood at (850) 644-2271.

If you have any questions or concerns regarding the study and would like to talk to someone other than the researchers, you are encouraged to contact the FSU IRB at telephone number 850-644-8633. You may also contact this office by email at <a href="https://humansubjects@fsu.edu">humansubjects@fsu.edu</a>, or by writing or in person at 2010 Levy Street, Research Building B, Suite 276, FSU Human Subjects Committee, Tallahassee, FL 32306-2742.

You will be given a copy of this form for your records.

#### **Statement of Consent**

| I have read the above information, I have consent to participate in this study. | ave asked questions and have received answers. I |
|---|---|
| Printed Name of Subject | _ |
| Signature of Subject | <br>Date |